CLINICAL TRIAL: NCT03304691
Title: The Molecular Basis of Erythrocyte Invasion by Plasmodium Vivax Into Duffy-Negative Erythrocytes in Mali
Brief Title: Molecular Basis of Erythrocyte Invasion by Plasmodium Vivax Into Duffy-Negative Erythrocytes in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917165; 17-I-N165
Record Dates: First submitted 2017-10-06; First posted 2017-10-09 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-02

CONDITIONS: Malaria
Keywords: Malaria; Parasitemia; Anemia; Ligand; Anopheles gambiae; Natural History
MeSH Terms: conditions — Malaria; Parasitemia; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bandiagara, Mali: Children of both sexes between 6 months and 10 years of age.
- Yirimadio, Bamako, Mali: Children and adults of both sexes 6 months and older.

SUMMARY:
Background:

Malaria is caused by parasites carried by some mosquitos. When the mosquitos bite people, the parasites can infect them. One of these parasites is Plasmodium vivax (P. vivax). Some children have P. vivax in their blood. They did not have malaria symptoms, but some also had a blood problem called anemia. This can make people feel tired or weak. This could have been caused by P. vivax. Researchers want to know how P. vivax infects these children, and if it affects their health.

Objective:

To collect blood, stool, and urine monthly from children to look for infections with P. vivax, worms, and other parasites.

Eligibility:

Children between 6 months and 10 years old

Design:

For screening, the study will be explained to the participant s parents or guardians, who will provide consent.

Participants will have a visit once a month for about 3 months, from November to January, and then for about 6 months from June to November 2018. Visits include:

Questions about their health

Medical history

Physical exam

Blood draw by pricking the finger tip

Urine and stool collection. They may collect these at home and bring them back.

If participants have P. vivax in their blood, them may need to come back to the clinic within 3 days. They will have blood taken from their arm using a needle.

If participants feel ill during the study, they can go to the clinic for an exam and blood tests.

If participants develop malaria while on the study, they will be treated.

Participants samples will be stored for future research studies.

...

DETAILED DESCRIPTION:
Plasmodium vivax was thought not to be a problem in Duffy blood group negative Africans. However, recent research has found that P. vivax infection occurs not only in areas where Duffy-positive and -negative people live side-by-side, but also in areas where populations are predominantly Duffy-negative, such as Bandiagara, Mali. In this region, our research group recently observed 25 P. vivax infections in children, all of whom were Duffy-negative. Furthermore, some preliminary data suggest that, despite having extremely low parasitemia and no malarial symptoms (no fever, muscle aches, or chills), the children of Bandiagara with P. vivax may have a drop in hemoglobin.

The present study involves two substudies to detect P. vivax infections in children and adults of two predominantly Duffy-negative Malian populations where P. vivax infections have previously been identified. The cohort study will be conducted in the Bandiagara region. We will conduct physical exams and collect blood, urine, and stool samples at baseline and monthly (urine samples will be collected only at baseline) for about 10 months. Our goal is to detect and characterize P. vivax infections, focusing on molecularly characterizing how P. vivax invades erythrocytes in Duffy-negative individuals. Specifically, we want to identify the parasite ligands involved in this invasion. We will use RNA sequencing (RNAseq) of P. vivax in blood samples of infected subjects to define the level of expression of parasite invasion ligands. From the parasite DNA found in blood samples, we will determine whether there is gene expansion of the parasite ligand Duffy binding protein (PvDBP) (the number of copies of PvDBP in each genome), and identify the sequence of PvDBP to determine whether it can bind an erythrocyte receptor other than the Duffy blood group antigen (i.e., Duffy-negative erythrocytes). An additional focus will be whether P. vivax leads to anemia in the Duffy-negative children.

In addition, we will conduct a cross-sectional study to investigate the prevalence of P. vivax in the general population in Yirimadio, a periurban setting of Bamako, which is the sole place in Mali besides Bandiagara where P. vivax infections have been reported in Duffy-negative individuals. This will be achieved by undertaking a cross-sectional survey. Subjects will provide blood for blood smear and filter paper analyses to identify the presence of P. vivax infection at 3 different time points.

ELIGIBILITY:
* INCLUSION CRITERIA:

For inclusion in the cohort substudy, a child must meet the following criteria:

1. Is greater than or equal to 6 months and less than or equal to 10 years of age
2. Residing in Bandiagara for at least 6 months prior to screening
3. Will be available to attend visits during this study
4. Agrees to provide urine and stool samples during this study
5. Agrees to allow storage of samples for future research.

For inclusion in the cross-sectional substudy, an individual must meet the following criteria:

1. Aged greater than or equal to 6 months;
2. Residing in Yirimadio for at least 6 months prior to screening.

EXCLUISION CRITERIA:

The following criterion is exclusionary in either substudy:

1) Has any underlying conditions that, in the judgement of the clinical investigators, could increase the risk to the subject.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be selected to enroll based on community permission and sensitization strategies for both the Bandiagara and Yirimadio sites.
Sampling Method: Non-Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Identify the P. vivax ligands for infection of Duffy blood group negative Africans by RNA sequencing (RNAseq) of blood from P. vivax cases. | Monthly surveillance visits throughout length of the study
  Identify the P. vivax ligands for infection of Duffy blood group negative Africans by RNA sequencing (RNAseq) of blood from P. vivax cases.

SECONDARY OUTCOMES:
Determine the prevalence of P. vivax in Yirimadio in Duffy negative population | Beginning, peak, and end of transmission season
Identify the vector populations in and around the study area that may transmit malaria, including during the dry season, as well as the infection rates in these populations. | Monthly surveillance visits throughout length of the study
Study the association between P. vivax parasitemia and anemia in Duffy-negative Africans. | Monthly surveillance visits throughout length of the study
Determine by stool examinations the presence of hypnozoites in the liver that fail to cause blood infections. | Monthly surveillance visits throughout length of the study
Determine the number of clones of P. vivax circulating in the community by DNA sequencing of polymorphic parasite proteins. | Monthly surveillance visits throughout length of the study

CONTACTS AND LOCATIONS:
Overall Officials: Louis H Miller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Mali (2):
  - Yirimadio Community Health Center, Bamako
  - Bandiagara Malaria Program (BMP) Clinic, Bandiagara

REFERENCES:
- [Background] Gunalan K, Niangaly A, Thera MA, Doumbo OK, Miller LH. Plasmodium vivax Infections of Duffy-Negative Erythrocytes: Historically Undetected or a Recent Adaptation? Trends Parasitol. 2018 May;34(5):420-429. doi: 10.1016/j.pt.2018.02.006. Epub 2018 Mar 9. PMID 29530446
- [Background] Gunalan K, Sa JM, Moraes Barros RR, Anzick SL, Caleon RL, Mershon JP, Kanakabandi K, Paneru M, Virtaneva K, Martens C, Barnwell JW, Ribeiro JM, Miller LH. Transcriptome profiling of Plasmodium vivax in Saimiri monkeys identifies potential ligands for invasion. Proc Natl Acad Sci U S A. 2019 Apr 2;116(14):7053-7061. doi: 10.1073/pnas.1818485116. Epub 2019 Mar 14. PMID 30872477
- [Background] Niangaly A, Karthigayan Gunalan, Amed Ouattara, Coulibaly D, Sa JM, Adams M, Travassos MA, Ferrero J, Laurens MB, Kone AK, Thera MA, Plowe CV, Miller LH, Doumbo OK. Plasmodium vivax Infections over 3 Years in Duffy Blood Group Negative Malians in Bandiagara, Mali. Am J Trop Med Hyg. 2017 Sep;97(3):744-752. doi: 10.4269/ajtmh.17-0254. Epub 2017 Jul 27. PMID 28749772